CLINICAL TRIAL: NCT02771158
Title: A Randomized Controlled Trial of Midodrine During Recovery Phase From Septic Shock
Brief Title: Midodrine During Recovery From Septic Shock
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study never started
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: temp-1187
Record Dates: First submitted 2016-03-28; First posted 2016-05-12 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Hypotension; Shock, Septic; Sepsis
Keywords: critical care; shock, septic; sepsis; hypotension; midodrine
MeSH Terms: conditions — Hypotension; Shock, Septic; Sepsis | interventions — Midodrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- midodrine (Experimental): randomization to midodrine 20 mg every 8 hours to be increased to a maximum of 40 mg every 8 hours until intravenous vasopressor discontinuation
  Interventions: Drug: Midodrine
- placebo (Placebo Comparator): randomization to placebo control
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Midodrine — midodrine is metabolized to an active metabolite, desglymidodrine, which is an alpha adrenergic antagonist that causes vasoconstriction of both venous and arterial vasculature, thereby increasing blood pressure
  Other Names: proamatine
  Arms: midodrine
Drug: placebo — placebo will be administered to double blind the study
  Arms: placebo

SUMMARY:
The purpose of this study is to determine whether midodrine administration decreases duration of intravenous vasopressors and intensive care unit length of stay for patients in septic shock.

ELIGIBILITY:
Inclusion Criteria:

* admitted to intensive care unit
* diagnosis of septic shock on intravenous vasopressors
* stable/decreasing doses of intravenous vasopressors
* stable/improving organ function

Exclusion Criteria:

* allergy to midodrine
* multiple intravenous vasopressors
* increasing intravenous vasopressor requirements
* worsening organ dysfunction
* severe bradycardia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-08 (Estimated); Primary Completion 2017-11-01 (Actual); Study Completion 2017-11-01 (Actual)

PRIMARY OUTCOMES:
duration of intravenous vasopressors | from enrollment until discontinuation of intravenous vasopressors, expected to be 3-5 days

SECONDARY OUTCOMES:
intensive care unit length of stay | from enrollment until eligible for discharge from intensive care unit, expected to be 4-7 days
re-institution of intravenous vasopressor | from enrollment until hospital discharge, expected to be up to 30 days
hospital length of stay | from enrollment until hospital discharge, expected to be up to 30 days
mortality | from enrollment until hospital discharge, expected to be up to 30 days
midodrine side effects requiring discontinuation | from enrollment until hospital discharge, expected to be up to 30 days
  including supine hypertension and bradycardia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Whitson MR, Mo E, Nabi T, Healy L, Koenig S, Narasimhan M, Mayo PH. Feasibility, Utility, and Safety of Midodrine During Recovery Phase From Septic Shock. Chest. 2016 Jun;149(6):1380-3. doi: 10.1016/j.chest.2016.02.657. Epub 2016 Mar 4. PMID 26953217